CLINICAL TRIAL: NCT01740167
Title: Health Promotion on Young Adults With High Risk Disability for Mental Health: Development and Evaluation of the Screen Prevention Model
Brief Title: Health Promotion on Young Adults With High Risk Disability for Mental Health
Acronym: HPMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NSC101-2511-S-039-003; DMR101-IRB2-222 (Other: ChinaMUH)
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Mental Health Wellness 1
Keywords: prodrome; mental illness; health promotion; lifestyle behavior
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle program (Experimental): health promotion lifestyle program : individual counseling, once a month, total 3 times.
  Interventions: Behavioral: health promotion lifestyle program

INTERVENTIONS:
Behavioral: health promotion lifestyle program — Individual counseling, once a month, total 3 times.

SUMMARY:
1. The positive outcomes reported by participants in experimental group after two weeks of interventions will be significantly better than before interventions.
2. The positive outcomes reported by participants in experimental group will be significantly better than those in control group after two weeks of providing prevention model interventions.
3. The positive outcomes reported by participants in experimental group will be significantly better than those in control group after six months of providing prevention model interventions.

DETAILED DESCRIPTION:
Early finding for people with high mental risk plays the important role in mental health promotion. In literature, before specific psychotic symptoms appear, individuals may experience a period of nonspecific symptoms and growing functional impairment. Early interventions may alter the natural course of mental diseases and improve treatment outcomes. So that, the purpose of this study is to develop a screen and prevention mode for identifying young adults with high risk status of mental health disability. The psychosocial intervention strategies for emotional and cognitive support in prevention model based on health promotion theory will be used for this study. Participants in this experimental design study will be randomly assigned into experimental and control groups. Four scales and objective physical assessments are used for evaluating study outcomes. The pre- and post-test will be held before and one week after prevention interventions. In addition, follow-ups will be included for understanding long-term outcomes of the effectiveness of the screen prevention model.

ELIGIBILITY:
Inclusion Criteria:

* age 20-65 years, (Chinese version of Schizotypal Personality Questionnaire-Brief > 17 scores, or Chinese Mandarin State Trait Anxiety Inventory Y2 > 60 scores), and agree to participants.

Exclusion Criteria:

* had been diagnosed as schizophrenia, bipolar disorders, and major depression.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Chinese version of Health-Promotion Lifestyle Profile-Short | 3 months

SECONDARY OUTCOMES:
Chinese version of Schizotypal Personality Questionnaire-Brief | 3 months

OTHER OUTCOMES:
Chinese mandarin version of State-Trait Anxiety Inventory from Y | 3 months
simple physical assessment | 3 months
Personal Inventory | 3 months
3 months physical activity assessment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Ma, PHD, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taiwan